CLINICAL TRIAL: NCT03475498
Title: A Major Determinant Focused on the ECG or Echocardiogram for Pacing-induced Cardiomyopathy (PICM) and Its Clinical Outcome (PICM Syndrome) : Prospective, Multi-center, Observational Cohort Study.
Brief Title: A Major Determinant Focused on the ECG or Echocardiogram for PICM and Its Clinical Outcome (PICM Syndrome)
Status: Recruiting | Type: Observational
Sponsor: Eulji University Hospital (Other)
Collaborators: Chungnam National University Hospital (Other); Chungbuk National University Hospital (Other); Dankook University (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Ki-Woon Kang, MD, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Other Study IDs: EMC 2018-01-013
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-05

CONDITIONS: Pacemaker Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Investigators exam to identify a biomarker (ECG or Echocardiogram parameter or genetic factor) as a determinant for occurrence of PICM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Chronic right ventricular pacing has a deleterious effect on left ventricular (LV) function, namely pacing-induced cardiomyopathy (PICM). Several parametes make difference of effect on the occurrence of PICM and its subsequent clinical outcomes. In particular, recognition of a major determinant focused on the ECG or echocardiographic parameters including strain or genetic factor for occurrence of PICM may lead to better identification of patients at high risk. Investigators prospectively enroll a participant with documented high risk of PICM and clinically follow-up to idenify clinical impact of PICM (PICM syndrome) over a long period of time.

DETAILED DESCRIPTION:
Investigators investigate a major determinant focused on the ECG or echocardiogram or genetic factor to predict the PICM after implantation of pacemaker. Not only QRS duration and mechanical strain but also genetic factor could be also investigated to predict the occurrence of PICM before diagnosis fo PICM

ELIGIBILITY:
Inclusion Criteria: mandatory (1 and 2) and optional (3 or 4)

1. Willng to participate in the study and able to sign informed consent
2. Undertaken ECG and echocardiogram including strain before and after device implantation

Exclusion Criteria:

1. Less than 18 years of age
2. Being pregnant or plan to become pregnant
3. Advanced heart failure waiting in heart transplantation
4. Have a life expectancy of less than 1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll at least 1000 device patients from multi-centers in order to identify and assess a determinant of PICM and its clinical outcomes (PICM syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Heart failure diagnosis and treatment | 5 years
  Occurrence of heart failure symptom, diagnosis and treatment

SECONDARY OUTCOMES:
Atrial and Ventricular arrhythmia diagnosis, heart failure admisssion and all-caused mortality | 5 years
  Occurrence of atrial, ventricular arrhythmia, hear failure admission and all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: KI-Woon Kang, MD PhD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (3):
- South Korea (3):
  - Chung-Buk University Hospital, Chungju
  - Chung-Nam University Hospital, Daejeon
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JH, Kang KW, Chin JY, Kim TS, Park JH, Choi YJ. Major determinant of the occurrence of pacing-induced cardiomyopathy in complete atrioventricular block: a multicentre, retrospective analysis over a 15-year period in South Korea. BMJ Open. 2018 Feb 8;8(2):e019048. doi: 10.1136/bmjopen-2017-019048. PMID 29439074
- [Background] Phung CD, Ezieme JA, Turrens JF. Hydrogen peroxide metabolism in skeletal muscle mitochondria. Arch Biochem Biophys. 1994 Dec;315(2):479-82. doi: 10.1006/abbi.1994.1528. PMID 7986095